CLINICAL TRIAL: NCT02042859
Title: Pilot Study to Assess Safety and Efficacy Of An Endoscopic Bipolar Radiofrequency Probe (EndoHPB) In the Management of Unresectable Bile Duct and Pancreatic Cancer
Brief Title: Radiofrequency Probe for Management of Unresectable Bile Duct and Pancreatic Cancer
Acronym: EndoHPB
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Ochsner Health System (Other)
Responsible Party: Principal Investigator, Virendra Joshi, Virendra Joshi, MD, Ochsner Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRFA
Record Dates: First submitted 2014-01-15; First posted 2014-01-23 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Pancreatic Cancer
Keywords: EndoHPB
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Endoscopic Bipolar RadioFrequency Probe used to remove tumors in bile duct to manage Pancreatic Cancer

SUMMARY:
The purpose of this study is to determine whether the use of an FDA approved endoscopic bipolar catheter (EndoHPB) will ablate tissue in malignant tumors within the pancreatic ducts.

DETAILED DESCRIPTION:
Only a small proportion of patients with biliary obstruction caused by cholangiocarcinoma or pancreatic cancer are suitable for surgical resection. Therefore most patients with malignant biliary obstruction will need palliation of their jaundice to relieve the symptoms of pruritus, malabsorption, sepsis and to minimize potential hepatorenal complications. Restoring biliary flow with relief of jaundice is the primary goal in the palliation of obstructive biliary malignancy. Drainage at endoscopic retrograde cholangiopancreatography (ECRP) is established as a safer approach than at percutaneous transhepatic cholangiography (PTC) because it has a lower risk of bile leak, infection and hemorrhage. ECRP is the first approach to relieve malignant biliary obstruction but sometimes it is not technically possible to stent the patient by this approach, then a PTC needs to be undertaken. Self expanding mesh metal stents (SEMS) were introduced back in the 1990s. Problems can still arise with the use of covered stents such as cholecystitis, pancreatitis or tumor overgrowth at the end of the stent, and not all studies have shown that covered stents actually reduce the problems of tumor ingrowth and consequent stent occlusion. EndoHPB can be deployed via an ERCP or PTC route. By using radiofrequency (RF) energy to heat the tissue in the duct prior to insertion of the stent, the surrounding tissue becomes coagulated and this may may delay tumor growth and the time before the stent lumen becomes blocked. Thereby this allows increased periods between the need for intervention and further stent deployment. If EndoHPB use of luminal RF is demonstrated to be effective in luminal tumor ablation, it may have an additional role as a form of neoadjuvant therapy in cholangiocarcinoma and pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Either gender greater than or equal to 18 years of age.
* Pancreatic Cancer or Cholangiocarcinoma unsuitable for surgical resection. Criteria of unresectability being based on 1) metastatic disease or 2) locally advanced disease.
* Biliary Obstruction
* Subjects capable of giving informed consent
* Life expectancy of at least 3 months

Exclusion Criteria:

* Cardiac Pacemaker
* Patient unstable for endoscopy
* Inability to give informed consent
* Uncorrected coagulopathy
* Pregnancy
* Karnofsky score less than 40%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Improvement in size(patency of bile duct) measured by cholangiography or cholangioscopy, immediately post ablation | Baseline through visit 7